CLINICAL TRIAL: NCT02976961
Title: A Personalized and Interactive Web-based Health Care Innovation to AdvanCe the QualIty of Life and CaRE of Patients with an Implantable Cardioverter Defibrillator
Brief Title: A Personalized and Interactive Web-based Health Care Innovation to Advance the Quality of Care
Acronym: ACQUIRE-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Schmidt Pedersen (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Susanne Schmidt Pedersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 31779
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Implantable Defibrillator User; Distress
Keywords: Information; Empowerment
MeSH Terms: conditions — Empowerment | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Implantable cardioverter defibrillator implant + usual care + supportive care given via an e-health platform. The supportive care consists of information, dialogue with a nurse or psychologist, CBT-based psychological intervention online, quizzes to increase knowledge
  Interventions: Other: Supportive care
- Usual care (No Intervention): Implantable cardioverter defibrillator implant + usual care

INTERVENTIONS:
Other: Supportive care — Information, guidance, supportive care, and psychological intervention
  Arms: Intervention

SUMMARY:
This study evaluates the clinical efficacy and cost-effectiveness of the ACQUIRE-ICD care innovation as add-on to usual care as compared to usual care alone in patients with an implantable cardioverter defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first-time ICD or CRT-D
* ≥18 years of age

Exclusion Criteria:

* Subcutaneous ICD
* Upgrade from a pacemaker to ICD or CRT
* History of psychiatric illness other than affective/anxiety disorders
* Cognitive impairments (e.g. dementia)
* Left ventricular assist device (LVAD) or upcoming LVAD implant
* Under evaluation or on the waiting list for heart transplantation
* No e-mail address
* Inability to manage or cope with computer technology
* Insufficient knowledge of the Danish language
* Participation in other randomized controlled trials unless of a technical nature
* Irresponsible to ask patient to participate according to GCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Device acceptance | 12 months
  Measured with the Florida Patient Acceptance Survey (FPAS)

SECONDARY OUTCOMES:
Health status (generic) | 12 and 24 months
  Measured with the Short Form Health Survey 12 items (SF-12)
Patient empowerment (ICD-EMPOWER) | 12 and 24 months
  Purpose-designed and disease-specific 14-item measure that measures patient empowerment
ICD patient concerns (ICDC) | 12 and 24 months
  8-item ICD Patients' Concern questionnaire that taps into fear of shock as reported by the patient
Symptoms of anxiety | 12 and 24 months
  Generalized Anxiety Disorder scale (GAD-7)
Symptoms of depression | 12 and 24 months
  Patient Health Questionnaire (PHQ-9)
Health status (heart failure specific) | 12 and 24 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Return to work | 12 and 24 months
  Purpose-designed questions
Time to first ICD therapy | 12 and 24 months
  Defined as ATP, cardioversion or shock
Time to first hospitalization due to a cardiac cause | 12 and 24 months
  Hospitalization due to a cardiac cause
Time to mortality | 12 and 24 months
  Mortality
Cost-effectiveness | 12 and 24 months
  Incremental cost gained per quality adjusted life year (QALY) and burden on health care professionals (physicians and nurses)). This will be measured with the EQ-5D-5L or captured from the patient's electronic health record (EHR; e.g. number of phone calls, emails, and consultations with patients), and purpose-designed questions.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne S Pedersen, PhD, Principal Investigator — University of Southern Denmark
Locations (5):
- Denmark (5):
  - Gentofte Hospital, Gentofte Municipality, Hellerup
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Zealand University Hospital - Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen SS, Skovbakke SJ, Wiil UK, Schmidt T, dePont Christensen R, Brandt CJ, Sorensen J, Vinther M, Larroude CE, Melchior TM, Riahi S, Smolderen KGE, Spertus JA, Johansen JB, Nielsen JC. Effectiveness of a comprehensive interactive eHealth intervention on patient-reported and clinical outcomes in patients with an implantable cardioverter defibrillator [ACQUIRE-ICD trial]: study protocol of a national Danish randomised controlled trial. BMC Cardiovasc Disord. 2018 Jul 3;18(1):136. doi: 10.1186/s12872-018-0872-7. PMID 29969990